CLINICAL TRIAL: NCT00611351
Title: Matched Unrelated Donor Allogeneic Hematopoietic Stem Cell Transplantation With a Conditioning Regimen of Targeted Busulfan, Cyclophosphamide, and Thymoglobulin
Brief Title: Busulfan, Cyclophosphamide, & Antithymocyte Globulin Followed by Stem Cell Transplant in Treating Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0122-05-FB; P30CA036727 (NIH)
Record Dates: First submitted 2008-02-07; First posted 2008-02-08 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Secondary Myelofibrosis
Keywords: graft versus host disease; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; untreated adult acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; stage III multiple myeloma; refractory multiple myeloma; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; secondary myelofibrosis; secondary acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent adult acute lymphoblastic leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult nasal type extranodal NK/T-cell lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; refractory hairy cell leukemia; stage I multiple myeloma; stage II multiple myeloma
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Extranodal NK-T-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Hairy Cell | interventions — Antilymphocyte Serum; Immunosuppressive Agents; Busulfan; Cyclophosphamide; Mycophenolic Acid; Tacrolimus; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Flow Cytometry; Pharmacogenomic Testing; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Unrelated Donor Allogeneic (Experimental): Matched unrelated donor allogeneic stem cell transplantation with a conditioning regimen of targeted busulfan, cyclophosphamide and thymoglobulin.
  Interventions: Biological: anti-thymocyte globulin; Drug: busulfan; Drug: cyclophosphamide; Drug: mycophenolate mofetil; Drug: tacrolimus; Genetic: polymerase chain reaction; Genetic: polymorphism analysis; Other: flow cytometry; Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
  Other Names: immunosuppressant
Drug: busulfan
  Other Names: Busulfex, Myleran
Drug: cyclophosphamide
  Other Names: cytophosphane
Drug: mycophenolate mofetil
  Other Names: CellCept
Drug: tacrolimus
  Other Names: Protopic, Envarsus XR, Astagraf XL
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: flow cytometry
Other: laboratory biomarker analysis
Other: pharmacogenomic studies
Other: pharmacological study
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor bone marrow transplant or peripheral stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When certain stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving busulfan together with cyclophosphamide and antithymocyte globulin followed by donor stem cell transplant works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the incidence of grade II-IV acute graft-versus-host disease in patients with hematologic cancer or other diseases treated with a myeloablative conditioning regimen comprising targeted (steady-state concentration of 800-1,000 ng/mL) busulfan, cyclophosphamide, and anti-thymocyte globulin followed by matched unrelated donor allogeneic hematopoietic stem cell transplantation.
* To determine the day +100 transplantation-related mortality in these patients.

Secondary

* To determine the effect of cyclophosphamide pharmacokinetic parameters on day +100 transplantation-related mortality in these patients.
* To determine the ability of low-dose anti-thymocyte globulin administered on day +5 to induce activation-induced cell death of activated donor lymphocytes.
* To determine the incidence of chronic graft-versus-host disease in patients treated with this regimen.
* To determine event-free and overall survival of patients treated with this regimen.
* To evaluate pharmacogenomic associations between genetic polymorphisms in drug disposition enzymes with the pharmacokinetics of busulfan and cyclophosphamide.

OUTLINE:

* Myeloablative conditioning regimen: Patients receive busulfan IV over 2 hours on days -8 to -5; cyclophosphamide IV over 4 hours on days -3 to -2; and anti-thymocyte globulin IV over 6 hours on day -3 and then over 4 hours on days -2, -1, and 5.
* Allogeneic hematopoietic stem cell transplantation: Patients undergo allogeneic bone marrow or peripheral blood stem cell infusion on day 0.
* Graft-versus-host-disease prophylaxis: Patients receive tacrolimus IV continuously or orally on days 6 to150, followed by an even taper to day 180 in the absence of graft-versus-host-disease. Patients also receive mycophenolate mofetil IV or orally beginning on day 6 and continuing to day 28.

Patients undergo blood collection periodically during study for pharmacokinetic, pharmacogenomic, and other translational studies. Genomic DNA extracted from blood samples is analyzed by polymerase chain reaction for genetic polymorphisms in cyclophosphamide/busulfan disposition enzymes. Activated donor lymphocytes are assessed using flow cytometry to measure activation-induced cell death, as reflected by apoptosis in activated T cells. Chimerism on or around day 100 is also assessed using fluorescence in situ hybridization analysis and DNA fingerprinting.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia
  * Acute lymphocytic leukemia
  * Chronic myelogenous leukemia beyond first chronic phase (i.e., 2nd chronic phase, accelerated phase, or blast crisis)
  * Multiple myeloma
  * Myelodysplastic syndromes
  * Malignant lymphoma
  * Myelofibrosis
* Requirement for myeloablative conditioning regimen confirmed by attending physician
* Available donor must meet the following criteria:

  * HLA phenotypically identical unrelated donor by low, intermediate, or high resolution for HLA class I antigens, and by high resolution for HLA class II antigens
  * Matched at the A, B, and DRβ1 loci
  * Single HLA-A or HLA-B antigen mismatch allowed
  * Meets all National Marrow Donor Program or foreign registry criteria for allogeneic bone marrow/stem cell donors
  * Peripheral blood stem cells are the preferred product on this study but bone marrow is allowed
* Karnofsky performance status 70-100%
* DLCO ≥ 50% predicted
* LVEF ≥ 45%
* Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 65 mL/min
* Serum total bilirubin ≤ 2.0 mg/dL
* Fertile patients must use effective contraception

Exclusion Criteria:

* No active uncontrolled infection
* Not pregnant or nursing/negative pregnancy test
* No HIV infection
* No chronic active hepatitis B or C or evidence of cirrhosis on liver biopsy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-06-07 (Actual); Primary Completion 2008-02-01 (Actual); Study Completion 2008-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Devetten, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unrelated Donor Allogeneic
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Unrelated Donor Allogeneic
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 50 [36 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5

OUTCOME MEASURES:

1. Primary Outcome: Transplantation-related Mortality at 100 Days Post-transplantation
Time Frame: at the 100 days post-transplant
Population: count of participants reflects number of participants not alive at 100 days post transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated Donor Allogeneic
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Incidence of Grade II-IV Acute Graft-versus-host-disease (GVHD)
Time Frame: at day 100 post transplantation
Population: count of participants represents number of participants with documented acute GVHD prior to day 100 post transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated Donor Allogeneic
Number analyzed (Participants) | 5
Participants | 4

3. Secondary Outcome: Overall Survival
Time Frame: 2 years post transplant
Population: Count of participants is the number of participant alive at the 2 year post transplant time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated Donor Allogeneic
Number analyzed (Participants) | 5
Participants | 2

4. Secondary Outcome: Event-free Survival
Time Frame: 2 years post transplant
Population: Number of participants at 2 years that experienced event-free survival.
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated Donor Allogeneic
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the time of consent until day plus 100 from transplant.
Description: Grade 4 anemia, thrombocytopenia, and leucopenia, grade 3 dysphagia, and grade 3 infertility are routinely expected for all patients participating in this protocol, so these events were not reported. Multiple grade 1 and grade 2 toxicities are also expected for all patients participating in this protocol; these events will not routinely be reported. All other toxicities > grade 3 will be reported.
Arm/Group | Unrelated Donor Allogeneic
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unrelated Donor Allogeneic (N=5)
Blood bilirubin increased (Investigations) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) — aspergillus pneumonia
Investigations - Other (Investigations) | 1 (1) — plasmacytoma
Infections and infestations - Other (Infections and infestations) | 1 (1) — positive blood culture
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unrelated Donor Allogeneic (N=5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 1 (1) — Epstein-Barr virus reactivation
Blood and lymphatic system - Other (Blood and lymphatic system disorders) | 1 (1) — hemorrhage
Blood bilirubin increased (Investigations) | 3 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Serum sickness (Immune system disorders) | 2 (2)
syncope (Nervous system disorders) | 1 (1)
Renal and Urinary disorders - Other (Renal and urinary disorders) | 2 (2) — renal failure
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1) — HHV-6
Seizure (Nervous system disorders) | 1 (1)
nervous system - Other (Nervous system disorders) | 1 (1) — mental status change related to seizure activity
Anorexia (Metabolism and nutrition disorders) | 1 (1)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
acute coronary syndrome (Cardiac disorders) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1) — septic emboli to brain
Endocarditis infective (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes